CLINICAL TRIAL: NCT03377296
Title: A Clinical Study to Assess the Safety of Controlled Human Plasmodium Vivax Malaria Infection Through Experimental Sporozoite Infection of Healthy Malaria-naïve UK Adults, and to Characterise Parasite Growth and Immune Responses to P.Vivax
Brief Title: Study of Controlled Human Plasmodium Vivax Infection
Acronym: VAC068
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAC068; 228948 (Other: IRAS)
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasmodium Vivax infection (Experimental): Both volunteers will be infected with Plasmodium Vivax (as described below in full in "Interventions"). i.e., there is only one arm to this study.
  Interventions: Other: Plasmodium vivax infection; Procedure: Collection of 250mL blood from each volunteer (N=2)

INTERVENTIONS:
Other: Plasmodium vivax infection — Two healthy human volunteers are exposed to the bites of five infectious mosquitoes per participant (by placing their forearms over the pot containing mosquitoes) for 5-10 minutes. Fed mosquitoes (as indicated by the presence of a blood meal in the abdomen) are individually dissected and assessed for sporozoite load (graded 0 to +4; a gland rating of +2 or more, representing 10 or more observed sporozoites, qualifies as being infectious). If, by this method the volunteer is found to have been inoculated by less than five infected mosquitoes, further mosquitoes are allowed to feed on the volunteer until a total of 5 appropriately infected mosquitoes have fed. The bite-challenge procedure continues until the subject has been bitten by 5 infectious mosquitoes.
Procedure: Collection of 250mL blood from each volunteer (N=2) — Collection of 250mL of P. vivax-infected blood from each volunteer when a threshold parasitaemia/ symptoms are met

SUMMARY:
This is a sporozoite-challenge clinical study with the primary aim of assessing the safety and feasibility of controlled human P. vivax malaria infection in two healthy volunteers. The investigators will also assess the growth of and the immune response to P. vivax infection, and assess the induction of sexual gametocytaemia post-CHMI via the natural route of malaria infection (mosquito bite). A secondary objective is to develop a blood inoculum of P. vivax-infected blood for future testing of candidate vaccines.

DETAILED DESCRIPTION:
This is a sporozoite-challenge clinical study with the primary aim of assessing the safety and feasibility of controlled human P. vivax malaria infection in two healthy volunteers. The investigators will also assess the growth of and the immune response to P. vivax infection, and assess the induction of sexual gametocytaemia post-CHMI via the natural route of malaria infection (mosquito bite). A secondary objective is to develop a blood inoculum of P. vivax-infected blood for future testing of candidate vaccines.

Two healthy, malaria-naïve adults aged between 18 and 50 years will be recruited at the CCVTM, Oxford. CHMI by sporozoites will be delivered by mosquito bite at Imperial College, London, and follow-up during the post-challenge period will be at the CCVTM in Oxford.

The two volunteers will have blood taken at regular intervals post-CHMI to assess the immune response to primary P. vivax infection, and also the gametocytaemia following P. vivax infection, and the volunteers will be monitored closely until the volunteers meet the criteria for treatment. Up to 250 mL (half a unit) of blood will be taken just prior to treatment from the two successfully infected volunteers (as determined by measurement of the parasitaemia) and frozen down for future use in blood-stage CHMI trials. The volunteers will be treated with a standard 60-hour course of oral artemether-lumefantrine (Riamet) followed by a 2-week course of partially-observed oral Primaquine for radical cure of P. vivax hypnozoites. The volunteers will be followed up for 3 months in the clinic and email follow-up will continue out to 5 years to monitor for clinical relapse.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy adult aged 18 to 50 years.

  * Blood group O, Rhesus negative.
  * Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
  * High metaboliser of primaquine (as determined by CYP2D6 genotype).
  * Normal serum levels of Glucose-6-phosphate dehydrogenase (G6PDH).
  * Satisfactory serum levels of Primaquine (when administered as test dose).
  * Able and willing (in the Investigator's opinion) to comply with all study requirements.
  * Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner.
  * Women only: Must practice continuous effective contraception* for the duration of the clinic visits (first 3 months post-CHMI).
  * Agreement to refrain from blood donation during the course of the study and for at least 5 years after the end of their involvement in the study.
  * Written informed consent to participate in the trial.
  * Reachable (24/7) by mobile phone during the period between CHMI and completion of all antimalarial treatment.
  * Willing to take a curative anti-malaria regimen following CHMI.
  * Willing to be admitted to the research bay on the John Warin ward at the Churchill Hospital for blood donation and clinical monitoring, until antimalarial treatment is underway and their symptoms are settling.
  * Willing to reside in Oxford for the duration of the study, until all antimalarials have been completed.
  * Answer all questions on the informed consent quiz correctly. * Female volunteers are required to use an effective form of contraception during the course of the study as malaria challenge could pose a serious risk to both maternal health and the unborn foetus.

Acceptable forms of contraception for female volunteers include:

* Established use of oral, injected or implanted hormonal methods of contraception (an additional form of contraception will be required when taking the antimalarial medication, as this can interfere with the efficacy of hormonal contraception).
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Total abdominal hysterectomy.
* Barrier methods of contraception (condom or occlusive cap with spermicide).
* Male sterilisation, if the vasectomised partner is the sole partner for the subject.
* True abstinence, when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

* • History of clinical malaria (any species).

  * Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
  * Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
  * Blood group A/B and/or Rhesus positive.
  * Red blood cells negative for the Duffy antigen/chemokine receptor (DARC).
  * Glucose-6-phosphate dehydrogenase (G6PDH) deficient.
  * Inadequate serum levels of Primaquine (when administered as test dose).
  * Current anaemia (Haemoglobin < 9 g/dL).
  * Use of immunoglobulins or blood products (e.g., blood transfusion) at any time in the past.
  * History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
  * Venepuncture unlikely to allow a 250 mL blood donation (as determined by the Investigator).
  * Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
  * Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
  * Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
  * History of allergic disease or reactions likely to be exacerbated by malaria infection.
  * Pregnancy, lactation or intention to become pregnant during the study.
  * Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
  * Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
  * Any clinical condition known to prolong the QT interval.
  * History of cardiac arrhythmia, including clinically relevant bradycardia.
  * Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
  * Family history of congenital QT prolongation or sudden death.
  * Contraindications to the use of both of the proposed anti-malarial medications; Riamet Malarone.
  * Contraindications to the use of Primaquine.
  * History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
  * History of serious psychiatric condition that may affect participation in the study.
  * Any other serious chronic illness requiring hospital specialist supervision.
  * Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 standard UK units every week.
  * Suspected or known injecting drug abuse in the 5 years preceding enrolment.
  * Hepatitis B surface antigen (HBsAg) detected in serum.
  * Seropositive for HTLV I or II (antibodies to HTLV) at screening.
  * Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
  * Seropositive for RPR (antibodies to syphilis) at screening.
  * Positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
  * Volunteers unable to be closely followed for social, geographic or psychological reasons.
  * Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in Appendix A.
  * Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Testing for HIV, HTLV, hepatitis B and C and syphilis will be performed at screening and then repeated 1 week prior to CHMI (day C-7) to ensure no new acquisition of infection prior to blood donation. Other infections will be screened for if the volunteer has recently travelled to an area where they may have been exposed to a blood-borne infection that could theoretically be transmitted to another healthy volunteer during a future blood-stage challenge.

- Exclusion criteria on day of CHMI

The following constitute absolute contraindications to CHMI:

* Acute disease, defined as moderate or severe illness with or without fever.
* Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of (Serious) Adverse Events following P. vivax CHMI | Up to 21 days post challenge
  Safety of P. vivax CHMI, as measured by incidence of (Serious) Adverse Events (Safety and Tolerability)
Clinical symptoms of malaria infection post CHMI | Up to 21 days post challenge
  Measure of successful infection (development of clinical symptoms of malaria)
Parasitaemia post CHMI | Up to 90 days post challenge
  Measure of successful infection (development of detectable persistent parasitaemia) symptoms).
Immune response to P. vivax | Up to 90 days post challlenge
  Immune response to P. vivax, as measured by antibody, B cell and T cell responses.
Gametocytaemia | Up to 90 days post challenge
  Gametocytaemia, as measured by qPCR

SECONDARY OUTCOMES:
Collection and freezing down of P. vivax-infected blood. | Collected between day 8 and day 14 post challenge, determined by symptoms and parasitaemia
  Collection and freezing down of up to 250 mL P. vivax-infected blood from 2 volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology & Tropical Medicine, Oxford, Oxfordshire
  - John Warin Ward, Oxford University NHS Foundation Trust, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Minassian AM, Themistocleous Y, Silk SE, Barrett JR, Kemp A, Quinkert D, Nielsen CM, Edwards NJ, Rawlinson TA, Ramos Lopez F, Roobsoong W, Ellis KJ, Cho JS, Aunin E, Otto TD, Reid AJ, Bach FA, Labbe GM, Poulton ID, Marini A, Zaric M, Mulatier M, Lopez Ramon R, Baker M, Mitton CH, Sousa JC, Rachaphaew N, Kumpitak C, Maneechai N, Suansomjit C, Piteekan T, Hou MM, Khozoee B, McHugh K, Roberts DJ, Lawrie AM, Blagborough AM, Nugent FL, Taylor IJ, Johnson KJ, Spence PJ, Sattabongkot J, Biswas S, Rayner JC, Draper SJ. Controlled human malaria infection with a clone of Plasmodium vivax with high-quality genome assembly. JCI Insight. 2021 Dec 8;6(23):e152465. doi: 10.1172/jci.insight.152465. PMID 34609964